CLINICAL TRIAL: NCT02466854
Title: Bleeding Complications in a Multicenter Registry of Patients Discharged With Diagnosis of Acute Coronary Syndrome and Underwent Percutaneous Coronary Intervention
Brief Title: Bleeding Complications in a Multicenter Registry of Patients Discharged With Diagnosis of Acute Coronary Syndrome
Acronym: BleeMACS
Status: Completed | Type: Observational
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, SERGIO RAPOSEIRAS ROUBÍN, MD, PhD, University of Santiago de Compostela
Other Study IDs: USantiago; Cardiochus (Registry Identifier: BleeMACS)
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Bleeding; Acute Coronary Syndrome; percutaneous coronary intervention; 1 year follow up
MeSH Terms: conditions — Acute Coronary Syndrome; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The BleeMACS (Bleeding complications in a Multicenter registry of patients discharged with diagnosis of Acute Coronary Syndrome) registry is an international observational database of bleeding outcomes for patients who are discharged with diagnosis of ACS and underwent Percutaneous Coronary Intervention (PCI), including myocardial infarction or unstable angina.

BleeMACS registry enrolls a total of more than 15,000 patients, including data from 16 hospitals in 11 countries: North America (Canada), South America (Brazil) Europe (Germany, Netherlands, Poland, Spain, Italy, Macedonia, Greece), and Asia (Japan and China).

The end-point of this study is to characterize patients at high risk of bleeding and to develop a risk score to accurately predict the risk of major bleeding within the first year after discharge from the hospital for an ACS.

DETAILED DESCRIPTION:
In December 2014, given the actual need for rigorous multicenter clinical investigation to test the safety of antithrombotic and contemporary therapies in patients with acute coronary syndromes (ACS), Dr. Sergio Raposeiras-Roubín and Dr. Emad Abu-Assi launched the BleeMACS (Bleeding complications in a Multicenter registry of patients discharged with diagnosis of Acute Coronary Syndrome) project.

Antithrombotic medication is commonly used for secondary prevention in patients following an ACS. This therapy, along with the invasive strategies, has been proved as effective, although it increases the risk of bleeding, which may counteract its benefits.

A growing body of evidence has demonstrated that the risk of death in patients with ACS is affected not only by recurrent ischemic events but also by major bleeding. Bleeding complications is the downside of antithrombotic therapy, as they were consistently associated with short- and long-term mortality, in addition to increase the risk of new thrombotic events particularly due to temporary or permanent modification/suspension of antithrombotic therapy, which is especially relevant in the first year after an ACS.

At present, there are several risk scores for predicting bleeding at short-term (during the hospitalization stage and at 30 days). However, at medium and long-term (i.e., ≤ 1 year), there is no available predicting systems to help clinicians quantify the bleeding risk of their patients. How could physicians predict the risk of bleeding after hospital discharge for ACS?

The purpose of this project was focused on helping clinicians to estimate the patient's baseline risk of major bleeding within the first year following an ACS. The investigators aim to identify the independent predictors of major bleeding at 1-year in order to develop a user-friendly bleeding risk score. The scoring system that the investigators intended to design using the data from the present registry would help clinicians in the decision-making process by identifying the optimal antithrombotic strategy, focusing closer attention to the patients with high risk of bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients discharged with diagnosis of an Acute Coronary Syndrome (ACS)
2. Undergoing percutaneous coronary intervention (PCI).
3. One year follow-up (except death)

Exclusion Criteria:

1. Patients who died during hospitalization.
2. Patients without coronary artery disease (basing on the definitions of criteria 2).
3. Patients who did not undergo PCI (simple balloon angioplasty, stent implantation and/or tromboaspiration).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients discharged with diagnosis of Acute Coronary Syndrome underwent percutaneous coronary intervention with at least 1 year of follow-up (except death)
Sampling Method: Probability Sample
Enrollment: 15401 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Serious bleeding | First year after discharge by acute coronary syndrome
  Bleeding requiring hospitalization and/or transfusion within the first year after hospital-discharge by acute coronary syndrome

CONTACTS AND LOCATIONS:
Overall Officials: SERGIO RAPOSEIRAS-ROUBIN, MD, PhD, Study Chair — University Clinical Hospital of Santiago de Compostela

REFERENCES:
- [Derived] Zheng W, Huang X, Wang X, Suo M, Yan Y, Gong W, Ai H, Que B, Nie S. Impact of multimorbidity patterns on outcomes and treatment in patients with coronary artery disease. Eur Heart J Open. 2024 Mar 27;4(2):oeae009. doi: 10.1093/ehjopen/oeae009. eCollection 2024 Mar. PMID 38544919
- [Derived] Zhang D, Gao H, Song X, Raposeiras-Roubin S, Abu-Assi E, Paulo Simao Henriques J, D'Ascenzo F, Saucedo J, Ramon Gonzalez-Juanatey J, Wilton SB, Kikkert WJ, Nunez-Gil I, Ariza-Sole A, Alexopoulos D, Liebetrau C, Kawaji T, Moretti C, Huczek Z, Nie S, Fujii T, Correia L, Kawashiri MA, Southern D, Kalpak O; Bleeding complications in a Multicenter registry of patients discharged with diagnosis of Acute Coronary Syndrome BleeMACS Registry Investigators. Optimal medical therapy improves outcomes in patients with diabetes mellitus and acute myocardial infarction. Diabetes Res Clin Pract. 2023 Sep;203:110833. doi: 10.1016/j.diabres.2023.110833. Epub 2023 Jul 20. PMID 37478977
- [Derived] Zhang D, Song X, Raposeiras-Roubin S, Abu-Assi E, Simao Henriques JP, D'Ascenzo F, Saucedo J, Gonzalez-Juanatey JR, Wilton SB, Kikkert WJ, Nunez-Gil I, Ariza-Sole A, Alexopoulos D, Liebetrau C, Kawaji T, Moretti C, Huczek Z, Nie S, Fujii T, Correia L, Kawashiri MA, Southern D, Kalpak O. Evaluation of optimal medical therapy in acute myocardial infarction patients with prior stroke. Ther Adv Chronic Dis. 2021 Sep 29;12:20406223211046999. doi: 10.1177/20406223211046999. eCollection 2021. PMID 34729148
- [Derived] Raposeiras-Roubin S, Faxen J, Iniguez-Romo A, Henriques JPS, D'Ascenzo F, Saucedo J, Szummer K, Jernberg T, James SK, Juanatey JRG, Wilton SB, Kikkert WJ, Nunez-Gil I, Ariza-Sole A, Song X, Alexopoulos D, Liebetrau C, Kawaji T, Moretti C, Huczek Z, Nie SP, Fujii T, Correia L, Kawashiri MA, Caneiro-Queija B, Cobas-Paz R, Acuna JMG, Southern D, Alfonso E, Terol B, Garay A, Zhang D, Chen Y, Xanthopoulou I, Osman N, Mollmann H, Shiomi H, Giordana F, Gaita F, Kowara M, Filipiak K, Wang X, Yan Y, Fan JY, Ikari Y, Nakahayshi T, Sakata K, Yamagishi M, Kalpak O, Kedev S, Rivera-Asenjo D, Abu-Assi E. Development and external validation of a post-discharge bleeding risk score in patients with acute coronary syndrome: The BleeMACS score. Int J Cardiol. 2018 Mar 1;254:10-15. doi: 10.1016/j.ijcard.2017.10.103. Epub 2018 Jan 28. PMID 29407077
- [Derived] Iannaccone M, D'Ascenzo F, Vadala P, Wilton SB, Noussan P, Colombo F, Raposeiras Roubin S, Abu Assi E, Gonzalez-Juanatey JR, Simao Henriques JP, Saucedo J, Kikkert WJ, Nunez-Gil I, Ariza-Sole A, Song XT, Alexopoulos D, Liebetrau C, Kawaji T, Moretti C, Garbo R, Huczek Z, Nie SP, Fujii T, Correia LC, Kawashiri MA, Garcia Acuna JM, Southern D, Alfonso E, Terol B, Garay A, Zhang D, Chen Y, Xanthopoulou I, Osman N, Mollmann H, Shiomi H, Giordana F, Kowara M, Filipiak K, Wang X, Yan Y, Fan JY, Ikari Y, Nakahashi T, Sakata K, Gaita F, Yamagishi M, Kalpak O, Kedev S. Prevalence and outcome of patients with cancer and acute coronary syndrome undergoing percutaneous coronary intervention: a BleeMACS substudy. Eur Heart J Acute Cardiovasc Care. 2018 Oct;7(7):631-638. doi: 10.1177/2048872617706501. Epub 2017 Jun 8. PMID 28593789
- [Derived] Iannaccone M, D Ascenzo F, De Filippo O, Gagliardi M, Southern DA, Raposeiras-Roubin S, Abu-Assi E, Henriques JPS, Saucedo J, Gonzalez-Juanatey JR, Wilton SB, Kikkert WJ, Nunez-Gil I, Ariza-Sole A, Song X, Alexopoulos D, Liebetrau C, Kawaji T, Huczek Z, Nie SP, Fujii T, Correia L, Kawashiri MA, Garcia-Acuna JM, Alfonso E, Terol B, Garay A, Zhang D, Chen Y, Xanthopoulou I, Osman N, Mollmann H, Shiomi H, Kowara M, Filipiak K, Wang X, Yan Y, Fan JY, Ikari Y, Nakahashi T, Sakata K, Yamagishi M, Moretti C, Gaita F, Kalpak O, Kedev S. Optimal Medical Therapy in Patients with Malignancy Undergoing Percutaneous Coronary Intervention for Acute Coronary Syndrome: a BleeMACS Sub-Study. Am J Cardiovasc Drugs. 2017 Feb;17(1):61-71. doi: 10.1007/s40256-016-0196-x. PMID 27738920